CLINICAL TRIAL: NCT06311149
Title: Multicenter Evaluation of Patients Using LATITUDE Monitoring System: Multitude Study
Brief Title: Multicenter Evaluation of Patients Using LATITUDE Monitoring System
Acronym: Multitude
Status: Recruiting | Type: Observational
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Sponsor
Other Study IDs: 479/2023/Oss/AOUFe
Record Dates: First submitted 2024-03-07; First posted 2024-03-15 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2023-12

CONDITIONS: Cardiovascular Diseases; Arrhythmias, Cardiac; Heart Failure; Sudden Cardiac Death
Keywords: Cardiac implantable electrical device; Implantable cardioverter defibrillator; Pacemaker; Cardiac resynchronization therapy; Subcutaneous defibrillator; Implantable cardiac monitor; Remote monitoring; Latitude monitoring system
MeSH Terms: conditions — Cardiovascular Diseases; Arrhythmias, Cardiac; Heart Failure; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Multitude is a registry of patients who receive commercially available CIEDs that remotely communicate through the LATITUDE monitoring system and transfer data to a central database.

The registry is designed to constitute a shared environment for the collection, management, analysis and reporting of clinical and diagnostic data, adopted by a network of European scientifically-motivated physicians who use rhythm management diagnostic and therapeutic solutions from Boston Scientific in their clinical practice.

The Multitude study will facilitate the sharing of scientific proposals within a large network of researchers, and it will allow researchers to record the experience with medical devices throughout the device and patient lifecycle.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing and capable of providing informed consent to collect/store/process personal health information by the sponsor or such consent is provided by a legally designated representative, if required by local law or regulation.
* Subject is:

  1. prospectively scheduled for receiving a device monitored through the LATITUDE monitoring system
  2. retrospectively enrolled after having received a device monitored through the LATITUDE monitoring system

Exclusion Criteria:

* Subject foreseen not to be followed at the enrolling center for at least 1 year after having received the device.
* Subject is receiving a device that is not approved for commercial use at the time of procedure.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The subjects will be recruited from the general patient population of the participating centers who are
  * receiving diagnosis or treatment using a device monitored through the LATITUDE monitoring system and
  * fulfilling all inclusion criteria and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2043-12-31 (Estimated); Study Completion 2043-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 10 years
  Mortality

SECONDARY OUTCOMES:
Hospitalization | 10 years
  Hospitalization
Device therapy | 10 years
  For therapeutic devices, e.g. ICDs, CRT-Ds, S-ICDs)
Device-related complications | 10 years
  Complication

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Bertini, Prof, Principal Investigator — Azienda Ospedaliera Universitaria di Ferrara
Locations (3):
- Italy (3):
  - Azienda Ospedaliero-Universitaria di Ferrara, Ferrara
  - Policlinico Federico II, Napoli
  - Ospedale "G.B. Grassi", Roma

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ferrick AM, Raj SR, Deneke T, Kojodjojo P, Lopez-Cabanillas N, Abe H, Boveda S, Chew DS, Choi JI, Dagres N, Dalal AS, Dechert BE, Frazier-Mills CG, Gilbert O, Han JK, Hewit S, Kneeland C, DeEllen Mirza S, Mittal S, Ricci RP, Runte M, Sinclair S, Alkmim-Teixeira R, Vandenberk B, Varma N. 2023 HRS/EHRA/APHRS/LAHRS expert consensus statement on practical management of the remote device clinic. Heart Rhythm. 2023 Sep;20(9):e92-e144. doi: 10.1016/j.hrthm.2023.03.1525. Epub 2023 May 19. PMID 37211145
- [Background] Glikson M, Nielsen JC, Kronborg MB, Michowitz Y, Auricchio A, Barbash IM, Barrabes JA, Boriani G, Braunschweig F, Brignole M, Burri H, Coats AJS, Deharo JC, Delgado V, Diller GP, Israel CW, Keren A, Knops RE, Kotecha D, Leclercq C, Merkely B, Starck C, Thylen I, Tolosana JM; ESC Scientific Document Group. 2021 ESC Guidelines on cardiac pacing and cardiac resynchronization therapy. Eur Heart J. 2021 Sep 14;42(35):3427-3520. doi: 10.1093/eurheartj/ehab364. No abstract available. PMID 34455430
- [Background] Zeppenfeld K, Tfelt-Hansen J, de Riva M, Winkel BG, Behr ER, Blom NA, Charron P, Corrado D, Dagres N, de Chillou C, Eckardt L, Friede T, Haugaa KH, Hocini M, Lambiase PD, Marijon E, Merino JL, Peichl P, Priori SG, Reichlin T, Schulz-Menger J, Sticherling C, Tzeis S, Verstrael A, Volterrani M; ESC Scientific Document Group. 2022 ESC Guidelines for the management of patients with ventricular arrhythmias and the prevention of sudden cardiac death. Eur Heart J. 2022 Oct 21;43(40):3997-4126. doi: 10.1093/eurheartj/ehac262. No abstract available. PMID 36017572
- [Background] Maines M, Tomasi G, Moggio P, Peruzza F, Catanzariti D, Angheben C, Simoncelli M, Degiampietro M, Piffer L, Valsecchi S, Del Greco M. Implementation of remote follow-up of cardiac implantable electronic devices in clinical practice: organizational implications and resource consumption. J Cardiovasc Med (Hagerstown). 2020 Sep;21(9):648-653. doi: 10.2459/JCM.0000000000001011. PMID 32628426
- [Background] Palmisano P, Melissano D, Zanotto G, Perego GB, Toselli T, Landolina M, Ricci RP; Italian Association of Arrhythmology, Cardiac Pacing (AIAC). Change in the use of remote monitoring of cardiac implantable electronic devices in Italian clinical practice over a 5-year period: results of two surveys promoted by the AIAC (Italian Association of Arrhythmology and Cardiac Pacing). J Cardiovasc Med (Hagerstown). 2020 Apr;21(4):305-314. doi: 10.2459/JCM.0000000000000950. PMID 32073430